CLINICAL TRIAL: NCT03569852
Title: The Effects of Four Weeks of Intermittent Fasting on Resting Energy Expenditure, Satiety Hormones, Body Composition, and Performance in Competitive Runners
Brief Title: Time Restricted Feeding in Male Runners
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: USDA, Western Human Nutrition Research Center (U.S. Federal Agency)
Collaborators: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: TRF 1223350
Record Dates: First submitted 2018-06-15; First posted 2018-06-26 (Actual); Last update posted 2020-04-01 (Actual); Status verified 2020-03

CONDITIONS: Fasting; Intermittent Fasting; Athletic Performance; Cardiovascular Risk Factor; Resting Energy Expenditure
MeSH Terms: conditions — Fasting; Intermittent Fasting

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group 1 (Experimental): Order of treatment, time restrictive feeding (16 hours fasting and 8 hours eating) followed by traditional eating pattern (12 hours fasted and 12 hours eating).
  Interventions: Behavioral: Time Restrictive Feeding; Behavioral: Traditional Eating Pattern
- Experimental Group 2 (Experimental): Order of treatment, traditional eating pattern (12 hours fasted and 12 hours eating) followed by time restrictive feeding (16 hours fasting and 8 hours eating).
  Interventions: Behavioral: Time Restrictive Feeding; Behavioral: Traditional Eating Pattern

INTERVENTIONS:
Behavioral: Time Restrictive Feeding — Volunteers will adhere to a form of time restrictive feeding, 16 hours fasting and 8 hours eating per day.
  Other Names: Intermittent Fasting
Behavioral: Traditional Eating Pattern — Volunteers will adhere to a more traditional eating pattern, 12 hours fasted and 12 hours eating per day.
  Other Names: Normal Diet

SUMMARY:
This is a cross-over intervention study designed to evaluate how four weeks of time restricted feeding (16 hours fasting and 8 hours feeding), compared to four weeks of a more traditional eating pattern (12 hours fasting and 12 hours feeding), affects resting energy expenditure, subjective and biochemical markers of satiety and hunger, body composition, cardiovascular health, substrate utilization and fitness in male competitive runners.

DETAILED DESCRIPTION:
Weight loss and improvements in body composition (increasing muscle mass and decreasing fat mass) are common goals for both dieters and athletes. Although a traditional method of achieving this has been accomplished through caloric restriction, an alternate method that is becoming increasingly popular is fasting. Fasting is described as the absence of food and/or calorie-containing beverage consumption for a period of time. The majority of people fast for 8-10 hours daily, which occurs during the overnight period when people are asleep Intermittent fasting, specifically time-restricted feeding (TRF), has recently gained popularity because it is a more sustainable means of practicing fasting and it has been shown to enhance the loss of fat mass with or without caloric restriction. It has also been shown to enhance overall health due to reports of reduced fasting glucose, insulin resistance, triglycerides, and reduced total and low-density lipoprotein (LDL) cholesterol levels in obese women. Despite its growing popularity among athletes, there is scarce research on how adhering to this type of diet pattern affects athletic performance and other biochemical markers related to health. The participants in this study will be randomly assigned to either a traditional (12/12) or a time restrictive (16/8) eating pattern in a crossover design. Each pattern will last for four weeks with a minimum two week washout in between, and the participants will consume the same calorie and macronutrient amounts based on recommendations made by the American College of Sports Medicine (ACSM) for both eating patterns. The 12/12 pattern will require subjects to consume 5 meals (breakfast, lunch, dinner, and two snacks) per day within a 12 hour period suggested to be around 8am, 10am, 12pm, 3pm, and 7pm. The 16/8 pattern will require subjects to consume 3 meals in an 8-hour period suggested to be around 12pm, 3pm, and 7pm. Subjects may only consume water, unsweetened coffee, or unsweetened tea (no artificial sweeteners) during their periods of fasting. Subjects will perform all exercise in the morning before 8 am in the fasted state. Subjects will visit the Western Human Nutrition Research Center (WHNRC) for test days at baseline (study day 1), after four weeks of the first dietary intervention (study day 28), and at the start (study day 43) and end of the second dietary intervention (study day 70), for a total of 4 test days over the duration of 10 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Competitive runners who have been actively training for 3 or more years
* Weigh a minimum of 110 lbs
* Training 4-6 times per week and run a minimum of 20 miles per week
* Competed in a race within past 12 months at a distance of 5 - 26.1 km
* Willing to repeat same monthly training protocol during two 4-week interventions
* VO2max range of 40-70 ml/kg/min

Exclusion Criteria:

* Smoker
* Take medications that have cardiovascular or metabolic effects
* Taking dietary supplements
* Following a restrictive diet including restricting calories or carbohydrates
* Evidence of an eating disorder
* Major injuries in past 3 months
* Chronic disease that affects bone health, metabolism or the cardiorespiratory system
* Present with any contra-indication to exercise testing (cardiovascular abnormalities) as evaluated by study physician

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2018-07-15 (Actual); Primary Completion 2020-03-24 (Actual); Study Completion 2020-03-24 (Actual)

PRIMARY OUTCOMES:
Change in resting energy expenditure | Study day 1, 28, 43 and 70
  Resting energy expenditure will be measured using a metabolic cart

SECONDARY OUTCOMES:
Change in body composition | Study day 1, 28, 43 and 70
  Body composition, including fat mass and lean body mass, will be measured by dual-energy x-ray absorptiometry (DEXA) and expressed in kilograms (kg).
Change in substrate utilization during exercise | Study day 1, 28, 43 and 70
  Carbohydrate and fat utilized for energy will be measured using a metabolic cart
Change in cardiovascular fitness | Study day 1, 28, 43 and 70
  Time to run a 10 kilometer time trial on a treadmill expressed in minutes
Change in perceived feelings of hunger and fullness | Study day 1, 28, 43 and 70
  Perceived hunger and fullness will be measured using a visual analog scale. Responses will be a mark on an unsegmented line from 0 or "not at all" to 5 or "extremely."
Change in glucagon, a biomarker of hunger and satiety | Study day 1, 28, 43 and 70
  Fasting plasma will be analyzed for glucagon (pmol/L) as measured by enzyme-linked immunoabsorbant assay
Change in leptin, a biomarker of hunger and satiety | Study day 1, 28, 43 and 70
  Fasting plasma will be analyzed for leptin (pmol/L) as measured by enzyme-linked immunoabsorbant assay
Change in ghrelin, a biomarker of hunger and satiety | Study day 1, 28, 43 and 70
  Fasting plasma will be analyzed for ghrelin (pmol/L) as measured by enzyme-linked immunoabsorbant assay
Change in insulin | Study day 1, 28, 43 and 70
  Fasting plasma will be analyzed for insulin (pmol/L) as measured by enzyme-linked immunoabsorbant assay
Change in total cholesterol, a biomarker of cardiovascular health | Study day 1, 28, 43 and 70
  Fasting serum will be analyzed for total cholesterol (mmol/L) by Piccolo analyzer
Change in HDL cholesterol, a biomarker of cardiovascular health | Study day 1, 28, 43 and 70
  Fasting serum will be analyzed for HDL cholesterol (mmol/L) by Piccolo analyzer
Change in LDL cholesterol, a biomarker of cardiovascular health | Study day 1, 28, 43 and 70
  Fasting serum will be analyzed for LDL cholesterol (mmol/L) by Piccolo analyzer
Change in very low-density lipoprotein (VLDL), a biomarker of cardiovascular health | Study day 1, 28, 43 and 70
  Fasting serum will be analyzed for very low-density lipoprotein (VLDL) cholesterol (mmol/L) by Piccolo analyzer
Change in triglycerides, a biomarker of cardiovascular health | Study day 1, 28, 43 and 70
  Fasting serum will be analyzed for triglycerides (mmol/L) by Piccolo analyzer
Change in alanine aminotransferase, a biomarker of cardiovascular health | Study day 1, 28, 43 and 70
  Fasting serum will be analyzed for alanine aminotransferase (IU/L) by Piccolo analyzer
Change in aspartate aminotransferase, a biomarker of cardiovascular health | Study day 1, 28, 43 and 70
  Fasting serum will be analyzed for aspartate aminotransferase (IU/L) by Piccolo analyzer
Change in glucose | Study day 1, 28, 43 and 70
  Fasting serum will be analyzed for glucose (mmol/L) by Piccolo analyzer

CONTACTS AND LOCATIONS:
Overall Officials: Gretchen Casazza, PhD, Principal Investigator — University of California, Davis
Locations (1):
- UC Davis, Western Human Nutrition Research Center, Davis, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Maughan RJ, Fallah J, Coyle EF. The effects of fasting on metabolism and performance. Br J Sports Med. 2010 Jun;44(7):490-4. doi: 10.1136/bjsm.2010.072181. Epub 2010 May 19. PMID 20484315
- [Background] Patterson RE, Sears DD. Metabolic Effects of Intermittent Fasting. Annu Rev Nutr. 2017 Aug 21;37:371-393. doi: 10.1146/annurev-nutr-071816-064634. Epub 2017 Jul 17. PMID 28715993
- [Background] Roy AS, Bandyopadhyay A. Effect of Ramadan intermittent fasting on selective fitness profile parameters in young untrained Muslim men. BMJ Open Sport Exerc Med. 2015 Sep 30;1(1):e000020. doi: 10.1136/bmjsem-2015-000020. eCollection 2015. PMID 27900122
- [Background] Tinsley GM, La Bounty PM. Effects of intermittent fasting on body composition and clinical health markers in humans. Nutr Rev. 2015 Oct;73(10):661-74. doi: 10.1093/nutrit/nuv041. Epub 2015 Sep 15. PMID 26374764
- [Background] Klempel MC, Kroeger CM, Bhutani S, Trepanowski JF, Varady KA. Intermittent fasting combined with calorie restriction is effective for weight loss and cardio-protection in obese women. Nutr J. 2012 Nov 21;11:98. doi: 10.1186/1475-2891-11-98. PMID 23171320
- [Background] Chaouachi A, Coutts AJ, Chamari K, Wong del P, Chaouachi M, Chtara M, Roky R, Amri M. Effect of Ramadan intermittent fasting on aerobic and anaerobic performance and perception of fatigue in male elite judo athletes. J Strength Cond Res. 2009 Dec;23(9):2702-9. doi: 10.1519/JSC.0b013e3181bc17fc. PMID 19910805
- [Background] Moro T, Tinsley G, Bianco A, Marcolin G, Pacelli QF, Battaglia G, Palma A, Gentil P, Neri M, Paoli A. Effects of eight weeks of time-restricted feeding (16/8) on basal metabolism, maximal strength, body composition, inflammation, and cardiovascular risk factors in resistance-trained males. J Transl Med. 2016 Oct 13;14(1):290. doi: 10.1186/s12967-016-1044-0. PMID 27737674
- [Background] Tinsley GM, Forsse JS, Butler NK, Paoli A, Bane AA, La Bounty PM, Morgan GB, Grandjean PW. Time-restricted feeding in young men performing resistance training: A randomized controlled trial. Eur J Sport Sci. 2017 Mar;17(2):200-207. doi: 10.1080/17461391.2016.1223173. Epub 2016 Aug 22. PMID 27550719
- [Background] Weigle DS, Duell PB, Connor WE, Steiner RA, Soules MR, Kuijper JL. Effect of fasting, refeeding, and dietary fat restriction on plasma leptin levels. J Clin Endocrinol Metab. 1997 Feb;82(2):561-5. doi: 10.1210/jcem.82.2.3757. PMID 9024254
- [Derived] Allaf M, Elghazaly H, Mohamed OG, Fareen MFK, Zaman S, Salmasi AM, Tsilidis K, Dehghan A. Intermittent fasting for the prevention of cardiovascular disease. Cochrane Database Syst Rev. 2021 Jan 29;1(1):CD013496. doi: 10.1002/14651858.CD013496.pub2. PMID 33512717